CLINICAL TRIAL: NCT01666327
Title: An Open-Label Study to Evaluate the Safety, Tolerability, Pharmacodynamics of a Single Oral Dose of MT-1303 in Subjects With Inflammatory Bowel Disease.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of MT-1303 in Subjects With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-E03
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — amiselimod

ARMS (1):
- MT-1303 (Experimental)
  Interventions: Drug: MT-1303

INTERVENTIONS:
Drug: MT-1303

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of a single oral dose of MT-1303 in subjects with inflammatory bowel disease.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, single-dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of MT-1303 in subjects with inflammatory bowel disease (Crohn's Disease and Ulcerative Colitis).

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) ranging from 16 to 34 kg/m2
* Subjects who were diagnosed as Crohn's Disease or Ulcerative Colitis at least 6 months prior to Screening, clinically confirmed either by radiological, endoscopic or histological examination.
* Subjects who have had at least one flare within 18 months prior to Screening.
* Confirmed medical records of inflammatory lesions in intestinal tract

Exclusion Criteria:

* Present or past history of clinically significant gastrointestinal surgery.
* Present or past history of clinically significant stenosis, stricture or fistula in small intestine or colon.
* Known hypersensitivity to any formulation excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose of MT-1303 assessed by number of participants with adverse events | 1month
Peak plasma concentration (Cmax) of MT-1303 and its metabolite | 15 time points up to 1 month
Area under the plasma concentration versus time curve (AUC) of MT-1303 and its metabolite | 15 time points up to 1 month

SECONDARY OUTCOMES:
Pharmacodynamic effect of MT-1303 on lymphocyte count | 16 time points up to 1 month
Exploratory parameter : C-reactive protein (CRP) | 4 time points up to 1 week
Exploratory parameter :Erythrocyte sedimentation (ESR) | 4 time points up to 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Nottingham, United Kingdom